CLINICAL TRIAL: NCT05337930
Title: 'Happyr Tracking': Feasibility of a Developmentally-tailored Mobile App for Tracking Mood and Pain in Children With Migraine
Brief Title: Feasibility of a Developmentally-tailored Mobile App for Tracking Mood and Pain in Children With Migraine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants enrolled in the study
Sponsor: Happyr Ltd (Industry)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 308617
Record Dates: First submitted 2022-03-29; First posted 2022-04-20 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2022-08

CONDITIONS: Primary Headache Disorder
Keywords: migraine; primary headache; tension type headache; pediatric headache; chronic pain
MeSH Terms: conditions — Headache Disorders, Primary; Migraine Disorders; Tension-Type Headache; Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other): Study participants will use the Happyr Health app, a mobile application to support CYP with primary headaches in coping with chronic pain, for eight weeks. For this study, a research version of the app will be provided via Google Play Store Testing Tracks and Apple TestFlight. In the app, a storyline and gamification elements engage CYP in filling out their headache diary and a regular mood diary.
  Interventions: Device: Happyr App

INTERVENTIONS:
Device: Happyr App — The Happyr app offers three main areas:
  (A) A mood diary in which a user can keep track of emotional wellbeing by answering three short questions.
  (B) A pain diary in which a user and supporter can record headache attacks by answering a set of predefined questions whenever a user experiences or has experienced a headache attack.
  (C) An overview section in which entries from the mood and pain diary are visualized for the user. In this section, a PDF document can also be exported with a summary of data from the symptom diary that can be taken to the clinician.
  A standardized notification is sent to each user at 6pm local time to remind them about logging their mood and symptoms of a headache attack.

SUMMARY:
This study aims to inform the continued development of a mobile app intended to support the treatment of CYP with migraine. After extensive public and patient involvement, Happyr Health has developed a mobile app that allows children and young people to track headache attacks and emotional wellbeing and to access coping techniques. With the use of gamification and storytelling elements, the app aims to engage children to be an active part in tracking and coping with their headaches. The outcomes of this study will inform future adaptations and development cycles of the Happyr Health app.

15 participants aged 10-16 will access the Happyr app for 8 weeks (= intervention). Primary outcomes of acceptability and implementation will be measured via surveys following the 8-week intervention in the app.

DETAILED DESCRIPTION:
The Happyr App is a mobile app to support children and young people with primary headaches in tracking their mood and symptoms. The app was developed in close collaboration with patients, their parents, and clinicians (pediatric neurologists, pediatric pain psychologists).

In the 'Happyr Tracking' study, we recruit 15 CYP aged 10-16 from the neurology department at Leeds Teaching Hospitals NHS Trust. Participants experience at least three primary headache attacks per month.

After receiving information on the study via the Principal Investigator (PI), those interested can contact the research team to receive access to the Happyr App.

In the app, participants and their parents/legal caregivers review information on the study and give their assent/consent. A copy of their signed assent/consent document will be sent to them as well as the research team and sponsor via email.

After creating their account, participants receive a survey in the app. As soon as completed, they can access the app's features. Participants are asked to make an entry to their mood diary at least once per day and to their pain diary only on days they experienced a pain attack. Participants are asked to send a PDF of their pain diary data (which they can export in the app) to the PI at the end of the intervention period (8 weeks).

After 8 weeks of using the app, participants will automatically receive another survey in the app to complete their participation. The pain diary export can be discussed with their clinician at their next appointment.

Outcomes of the study will be analyzed from the two in-app survey at beginning and end of the intervention period as well as usage data from the app analytics. The study objective is to understand the acceptability and feasibility of the Happyr App.

ELIGIBILITY:
Inclusion Criteria:

* With recurrent headaches (at least 3x per month)
* Access to a device (Android or iOS smartphone)
* Access to internet connection
* English-speaking

Exclusion Criteria:

* Secondary headaches
* Continuous headache
* Severe cognitive impairments
* Major comorbid medical or psychiatric illnesses (e.g. severe anxiety disorder)

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Acceptability Modified 'The mHealth App Usability Questionnaire (MAUQ)' | Post 8-week intervention
  Acceptability of the app to patients will be measured using items adapted from the mHealth App Usability Questionnaire. Questions use a Likert agreement response scale. A higher total score reflects greater acceptability (1 = strongly disagree (worse outcome); 5 = strongly agree (better outcome)). Our selected threshold for defining adequate acceptability is that 80% of participants will have an average score of at least 4/5 on the acceptability questionnaire (indicating moderate to high satisfaction with the app). Participants also will be asked in an open-ended item to provide general comments about their experience with the app.
Implementation (App usage frequency) | Post 8-week intervention
  Implementation will be evaluated using app analytics to measure the frequency of making a mood diary entry per week. Our selected threshold for defining acceptable implementation is that 80% of participants will submit an average of at least 4 completed daily diaries per week over the course of 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Munni Ray, Principal Investigator — The Leeds Teaching Hospitals NHS Trust
Locations (1):
- The Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom